CLINICAL TRIAL: NCT02052934
Title: A Phase 1 Dose Escalating Study of Double Mutant Heat-Labile Toxin LTR192G/L211A (dmLT) From Enterotoxigenic Escherichia Coli (ETEC) by Sublingual or Oral Immunization to Determine Safety and Immunogenicity of a Multi-dose Regimen in Adult Humans
Brief Title: Safety of Sublingual dmLT for ETEC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 12-0023; HHSN272201300016I
Record Dates: First submitted 2014-01-30; First posted 2014-02-03 (Estimated); Last update posted 2019-01-28 (Actual); Status verified 2016-12-07

CONDITIONS: Gastroenteritis Escherichia Coli
Keywords: Escherichia coli Infections; ETEC Candidate Vaccine; Immunogenicity
MeSH Terms: conditions — Escherichia coli Infections | interventions — Vaccines

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Cohort 1 (Experimental): Three sublingual (SL) doses of dMLT, 1 microgram (mcg), on Days 1, 15 and 29, 8 subjects
  Interventions: Biological: Recombinant Double Mutant Heat-Labile Toxin LT(R192G/L211A) (dmLT) Oral enterotoxigenic Escherichia coli (ETEC) Vaccine
- Cohort 2 (Experimental): Three SL doses of dMLT, 5 mcg, on Days 1, 15 and 29, 8 subjects
  Interventions: Biological: Recombinant Double Mutant Heat-Labile Toxin LT(R192G/L211A) (dmLT) Oral enterotoxigenic Escherichia coli (ETEC) Vaccine
- Cohort 3 (Experimental): Three SL doses of dMLT, 25 mcg, on Days 1, 15 and 29, 11 subjects
  Interventions: Biological: Recombinant Double Mutant Heat-Labile Toxin LT(R192G/L211A) (dmLT) Oral enterotoxigenic Escherichia coli (ETEC) Vaccine
- Cohort 4 (Experimental): Three SL doses of dMLT, 50 mcg, on Days 1, 15 and 29, 11 subjects
  Interventions: Biological: Recombinant Double Mutant Heat-Labile Toxin LT(R192G/L211A) (dmLT) Oral enterotoxigenic Escherichia coli (ETEC) Vaccine
- Cohort 5a (Experimental): Three SL doses of dMLT,25 mcg on Days 1, 15 and 29, 13 subjects.
  Interventions: Biological: Recombinant Double Mutant Heat-Labile Toxin LT(R192G/L211A) (dmLT) Oral enterotoxigenic Escherichia coli (ETEC) Vaccine
- Cohort 5b (Experimental): Three oral doses of dMLT, 25 mcg on Days 1, 15and 29, 13 subjects
  Interventions: Biological: Recombinant Double Mutant Heat-Labile Toxin LT(R192G/L211A) (dmLT) Oral enterotoxigenic Escherichia coli (ETEC) Vaccine

INTERVENTIONS:
Biological: Recombinant Double Mutant Heat-Labile Toxin LT(R192G/L211A) (dmLT) Oral enterotoxigenic Escherichia coli (ETEC) Vaccine — Attenuated, Recombinant Double Mutant Heat-Labile Toxin (dmLT) from Enterotoxigenic Escherichia coli (ETEC), LT(R192G/L211A); lot 1575. Subjects in 5 cohorts receive 3 doses ranging from 1 mcg to 50 mcg.
  Arms: Cohort 1; Cohort 2; Cohort 3; Cohort 4; Cohort 5a
Biological: Recombinant Double Mutant Heat-Labile Toxin LT(R192G/L211A) (dmLT) Oral enterotoxigenic Escherichia coli (ETEC) Vaccine — Attenuated, Recombinant Double Mutant Heat-Labile Toxin (dmLT) from Enterotoxigenic Escherichia coli (ETEC), LT(R192G/L211A); lot 1575. Subjects in 5b cohort receive 3 doses of 25 mcg.
  Arms: Cohort 5b

SUMMARY:
A Phase 1 dose escalating study of ETEC candidate vaccine to determine safety and immunogenicity of a multi-dose regimen in healthy adult volunteers. The study will be conducted at Cincinnati Children's Hospital Medical Center (CCHMC). The primary objectives assess the safety and tolerability of dmLT vaccine when administered in three doses sublingually over a range of dosages in healthy adult subjects. The secondary objectives assess long-term safety follow-up from immunization through Month 7 post vaccination, following three SL doses of dmLT vaccine over a range of dosages and comparing with three doses of a comparable dosage of oral vaccine. The study subject population is 52 healthy adult male and female subjects, ages 18 to 45. Subject participation duration is approximately 8 months with study duration of approximately 1.5-2 years, including 6-7 months of follow-up.

DETAILED DESCRIPTION:
Despite the public health burden of Enterotoxigenic Escherichia coli (ETEC) on travelers, deployed soldiers and, most significantly, young children in the developing world, there is no licensed vaccine against ETEC enteritis.This is a Phase 1 study in healthy adults to determine the safety and immunogenicity of an ETEC candidate vaccine, attenuated recombinant dmLT from ETEC, administered by the SL (Sublingual) or Oral Immunization. The study subject population is 52 healthy adult male and female subjects, ages 18 to 45. Subject participation duration is approximately 8 months with study duration of approximately 1.5-2 years, including 6-7 months of follow-up. Potential risks include subjects could develop varying degrees of diarrhea or other gastrointestinal symptoms (such as nausea, abdominal pain or cramping, gas, and decreased appetite). Blood drawing may be associated with pain and bruising at the site and rarely, with fainting or seizure. There is no direct benefit to subjects from participating in this study but the potential benefits to children and adults who may receive a future beneficial vaccine based on the results of this trial justify the more than minimal risk of the subjects who will participate in this trial. The primary objective is to assess the safety and tolerability of dmLT vaccine when administered in three doses sublingually over a range of dosages in healthy adult subjects. The secondary objectives are to assess long-term safety follow-up from immunization through Month 7 post vaccination, and following three SL doses of dmLT vaccine over a range of dosages and comparing with three doses of a comparable dosage of oral vaccine.

ELIGIBILITY:
Inclusion Criteria:

- Male or female ages 18-45, inclusive. - Provide written informed consent before initiation of any study procedures. - General good health, without (a) significant medical illness, (b) clinically significant physical examination findings, including vitals, as determined by the PI, and (c) screening laboratory values outside the site's normal limits. - Within 46 days of vaccination, have normal screening laboratories, per Appendix B for white blood cells (WBCs), hemoglobin (Hgb), platelets, absolute neutrophil count (ANC), sodium, potassium, chloride, bicarbonate, blood urea nitrogen (BUN), creatinine, alanine aminotransferase (ALT), aspartate aminotransferase (AST). - Have normal screening laboratories for urine protein Trace protein is acceptable. - HgbA1C <6.5% at screening. - Demonstrate comprehension of the protocol procedures and knowledge of study by passing a written examination (passing grade is at least 70 percent). - Agrees to complete all study visits and procedures. - Female subjects must be of non-childbearing potential (as defined as surgically sterile or postmenopausal for more than 1 year), or if of childbearing potential, must be using an effective method of birth control (e.g., use hormonal or barrier birth control such as implants, injectables, combined oral contraceptives, some intrauterine devices [IUDs], cervical sponges, diaphragms, condoms with spermicidal agents must have a vasectomized partner) within 2 months of vaccination, or practice abstinence and must agree to continue such precautions during the study and for 30 days after the Day 29 study visit. Male subjects must agree not to father a child for 30 days after the Day 29 study visit. A woman is eligible if she is monogamous with a vasectomized male. - Agrees not to participate in another clinical trial during the study period. - Agrees not to donate blood to a blood bank for 12 months after receiving the vaccine. - Potential subjects must be willing to adhere to the following prohibitions and restrictions during the course of the study to be eligible for participation: - Strenuous exercise (e.g., long distance running > 5km/day, weight lifting, or any physical activity to which the subject is not accustomed) is to be avoided during the overnight stay and for at least 72 hours prior to each study drug administration (and the Follow-up visit). - Subjects should not have donated blood in the 8 weeks prior to study entry.

Exclusion Criteria:

- Women who are pregnant or lactating or have a positive serum pregnancy test at screening or positive urine pregnancy test prior to vaccination. - Abnormal vital signs, defined as: -- Hypertension (systolic blood pressure >140 mm Hg or diastolic blood pressure >90 mm Hg) at rest on 2 separate days; or -- Palpated heart rate <55 or >100 beats/minute at rest on 2 separate days*; or *If heart rate between 45 and 55, subjects may be enrolled with an EKG that demonstrates normal sinus rhythm and does not document conduction disorders. --Temperature >/= 38.0 degrees C (100.4 degrees F) - Symptoms of an acute self-limited illness, including a temperature >/= 38.0 degrees C (100.4 degrees F), such as an upper respiratory infection or gastroenteritis within 7 days of administration of dmLT. - Positive hepatitis C, or HIV serology or positive hepatitis B serology not consistent with prior hepatitis B immunization. - Have a positive urine drug screen for opiates. - Subjects who are unwilling or unable to cease smoking for the duration of the overnight stay. - History of antimicrobial treatment in the 2 weeks before administration of dmLT. - Received previous experimental E. coli, LT, or cholera vaccines or live E. coli or Vibrio cholera challenges; or previous infection with cholera or diarrheagenic E. coli. - Abnormal routine bowel habits as defined by fewer than three stools per week or more than two stools per day in the past 6 months. - History of chronic gastrointestinal illness, including severe dyspepsia (mild or moderate heartburn or epigastric pain occurring no more than three times per week is permitted), or other significant gastrointestinal tract disease. - Regular use (weekly or more often) of laxatives, anti-diarrheal, anti-constipation, or antacid therapy. - History of major gastrointestinal surgery, excluding uncomplicated appendectomy or cholecystectomy. - Long-term use, defined as longer than 14 days, of oral steroids, parenteral steroids, or high-dose inhaled steroids (>800 mcg/day of beclomethasone dipropionate or equivalent) within the preceding 6 months. (Nasal and topical steroids are allowed). - Have a diagnosis of schizophrenia or other major psychiatric diagnosis. - Are receiving the following psychiatric drugs: aripiprazole, clozapine, ziprasidone, haloperidol, molindone, loxapine, thioridazine, thiothixene, pimozide, fluphenazine, risperidone, mesoridazine, quetiapine, trifluoperazine, chlorprothixene, chlorpromazine, perphenazine, trifluopromazine, olanzapine, carbamazepine, divalproex sodium, lithium carbonate, or lithium citrate. NOTE: Subjects who are receiving a single antidepressant drug and are stable for at least 3 months before enrollment without de-compensating symptoms are allowed to be enrolled in the study. - History of receiving Ig or other blood product within the 3 months before enrollment in this study. - Traveled to ETEC-endemic areas, defined as Africa, Middle East, South Asia, or Central or South America within the past 3 years or raised in a cholera or ETEC endemic area. - Received any licensed vaccine within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) before enrollment in this study or plans to receive any licensed vaccine within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) after any study vaccination. - An acute or chronic medical condition that, in the opinion of the investigator, would render administration of dmLT unsafe or would interfere with the evaluation of responses. This includes, but is not limited to: known or suspected immunodeficiency, known chronic liver disease, significant renal disease, unstable or pr ogressive neurological disorders, history of diabetes, cancer (other than a healed skin lesion), heart disease (in the hospital for a heart attack, history of irregular heart beat or fainting caused by an irregular heartbeat), unconsciousness (other than a single brief "concussion"), seizures (other than with fever when subject was a child <5 years old), asthma requiring treatment with inhaler or medication in the prior 2 years, autoimmune disease or eating disorder, and transplant recipients. - Received an experimental agent (vaccine, drug, biologic, device, blood product, or medication) within 1 month before enrollment in this study or expects to receive an experimental agent during the study. - History of alcohol or drug abuse in the last 5 years. - Plans to travel outside of the USA in the time between study vaccination and 28 days following the final vaccination. - Unable to spend up to 48 hours at an overnight facility following the administration of Dose 1. - Any condition that would, in the opinion of the Site Investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol. - Use of prescription or over-the-counter (OTC) medications that contain acetaminophen, aspirin, ibuprofen, and other non-steroidal anti-inflammatory drugs within 48 hours prior to receiving the investigational product. - Use of prescription acid suppression medication or OTC antacids within 72 hours of investigational product administration. - Subjects with autoimmune disorders, chronic inflammatory disorders or neurological disorders with a potential autoimmune correlation. - Subjects who planned to travel to an ETEC-endemic area, defined as Africa, Middle East, South Asia, or Central or South America, during the long-term safety follow-up period (6 months) of the study. - Known allergies to study compound. - Special populations, e.g., non-English speakers, children, illiterate or non-writing individuals, vulnerable populations. - Any abnormality of the palate.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2014-03-10 (Actual); Primary Completion 2016-11-02 (Actual); Study Completion 2016-11-02 (Actual)

PRIMARY OUTCOMES:
Occurrence of solicited reactogenic side effects through Day 8 following each vaccination. | Day 0 to Day 8
Occurrence of vaccine-related, non-solicited adverse events (AEs) for facial nerve disturbance through 75 days post third vaccination. | Day 29 through Day 104
Occurrence of vaccine-related, non-solicited adverse events (AEs) through Day 36 following first vaccination. | Day 0 to Day 36

SECONDARY OUTCOMES:
Occurrence of vaccine-related serious adverse events (SAEs) through 7 months following first vaccination. | Day 0 through Day 210
Proportion of subjects with =4-fold rise from the baseline in LT toxin neutralization titers. | Days 0, 8, 15, 22, 29, 36, 64 and 85
Proportion of subjects with >/= 2-fold rise from the baseline in dmLT-specific IgA- and IgG-ALS at any time after vaccination. | Days 0, 8, 15, 22, 29, 36, 64, and 85
Proportion of subjects with >/= 4-fold rise from the baseline in dmLT-specific fecal IgA or >/= 4-fold rise for the ratio of specific over total IgA after vaccination. | Days 0, 8, 15, 22, 29, 36, and 64
Proportion of subjects with >/= 4-fold rise from the baseline in dmLT-specific IgA- and IgG-ALS after vaccination. | Days 0, 8, 15, 20, 22, 29, 34, and 36
Proportion of subjects with >/= 4-fold rise from the baseline in dmLT-specific saliva IgA or >/= 4-fold rise for the ratio of specific over total IgA after vaccination. | Days 0, 8, 15, 22, 29, 36, and 64
Proportion of subjects with >/= 4-fold rise from the baseline in dmLT-specific serum IgA or IgG at any time after vaccination. | Days 0, 8, 15, 22, 29, 36, 64, and 85
Proportion of subjects with >8 IgA- or IgG-ASC/10^6 peripheral blood mononuclear cells (PBMCs) after vaccination. | Days 0, 8, 15, 20, 22, 29, 34, and 36
Proportion of subjects with IgG and IgA dmLT-specific circulating ASC expressing gut homing receptors. | Days 0 8, 15, 20, 22, 29, 34, and 36

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center - Gastroenterology, Hepatology and Nutrition, Cincinnati, Ohio, United States